CLINICAL TRIAL: NCT06207734
Title: Discontinuation of CDK4/6 Inhibitors in Patients With Metastatic HR Positive, HER2 Negative Breast Cancer With Durable Disease Control: A Randomized Low-intervention Phase II Trial of the AIO Working Groups Breast Cancer and Quality of Life
Brief Title: Discontinuation of CDK4/6 Inhibitors in Patients With Metastatic HR Positive, HER2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISCUSS
Record Dates: First submitted 2024-01-03; First posted 2024-01-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Metastatic HR positive, HER2 negative breast cancer; CDK4/6 inhibitors; Endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm CDK4/6 continuation (Active Comparator): * Continuation of CDK4/6 inhibitor treatment
  * Continuation of endocrine treatment
  Interventions: Drug: Continuation of CDK4/6 inhibitor Palbociclib; Drug: Continuation of CDK4/6 inhibitor -Palbociclib; Drug: Continuation of CDK4/6 inhibitor Abemaciclib
- Experimental arm CDK4/6 inhibitor discontinuation (Experimental): * Discontinuation of CDK4/6 inhibitor treatment
  * Continuation of endocrine treatment
  Interventions: Drug: Discontinuation of CDK4/6 inhibitor Palbociclib; Drug: Discontinuation of CDK4/6 inhibitor -Palbociclib; Drug: Discontinuation of CDK4/6 inhibitor Abemaciclib

INTERVENTIONS:
Drug: Continuation of CDK4/6 inhibitor Palbociclib — Continuation of CDK4/6 inhibitor Palbociclib
  Other Names: Study treatment
  Arms: Control arm CDK4/6 continuation
Drug: Discontinuation of CDK4/6 inhibitor Palbociclib — Discontinuation of CDK4/6 inhibitor Palbociclib
  Other Names: Study treatment
  Arms: Experimental arm CDK4/6 inhibitor discontinuation
Drug: Continuation of CDK4/6 inhibitor -Palbociclib — Continuation of CDK4/6 inhibitor -Palbociclib
  Other Names: Study treatment
  Arms: Control arm CDK4/6 continuation
Drug: Discontinuation of CDK4/6 inhibitor -Palbociclib — Discontinuation of CDK4/6 inhibitor -Palbociclib
  Other Names: Study treatment
  Arms: Experimental arm CDK4/6 inhibitor discontinuation
Drug: Continuation of CDK4/6 inhibitor Abemaciclib — Continuation of CDK4/6 inhibitor Abemaciclib
  Other Names: Study treatment
  Arms: Control arm CDK4/6 continuation
Drug: Discontinuation of CDK4/6 inhibitor Abemaciclib — Discontinuation of CDK4/6 inhibitor Abemaciclib
  Other Names: Study treatment
  Arms: Experimental arm CDK4/6 inhibitor discontinuation

SUMMARY:
This is a low-intervention, randomized, non-comparative, open-label, multicenter, prospective, phase II trial investigating discontinuation of CDK4/6 inhibitors in patients with metastatic HR positive, HER2 negative breast cancer with durable disease control.

DETAILED DESCRIPTION:
The primary objective is to evaluate long-term disease stabilization of CDK4/6 inhibitors discontinuation after a prolonged treatment period with continued endocrine therapy in breast cancer patients exhibiting at least stable disease after at least 12 months of combination treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient has given written informed consent
2. Patient is ≥ 18 years of age at time of signing the written informed consent
3. Patient has been diagnosed with histologically confirmed metastatic adenocarcinoma of the breast
4. Patient has documented histological or cytological confirmation of estrogen receptor positive (ER+) and HER2 negative (HER2-) disease
5. Patient has no curative treatment option by surgery or radiotherapy
6. Patient was treated with CDK4/6 inhibitor plus endocrine therapy for at least 12 months with disease control (complete remission, partial remission or stable disease) as judged by the treating physician before planned study treatment initiation
7. Patient has a preserved performance status (ECOG ≤ 2)
8. Patient has adequate bone marrow, renal and hepatic function:

   1. Hemoglobin > 9.0 g/dL
   2. Absolute neutrophil count judged as appropriate for study therapy by the investigator
   3. Platelets ≥ 100 x 109/L
   4. Calculated creatinine clearance judged as appropriate for study therapy by the investigator
   5. AST (SGOT) / ALT (SGPT) and alkaline phosphatase ≤ 2.5x ULN
   6. Serum albumin > 30 g/L
9. Patients considered postmenopausal according to one of the following definition:

   1. Women <50 years of age who are amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and whose levels of luteinizing hormone and follicle-stimulating hormone are in the post-menopausal institutional range
   2. Women ≥50 years of age who are amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago or had chemotherapy-induced menopause with last menses >1 year ago
   3. Artificially induced postmenopausal women (by Gonadotropin-releasing hormone [GnRH] analogs)
10. WOCBP must have a negative serum pregnancy test within 7 days prior to start of trial

Exclusion Criteria:

1. Patient has active (or history of) brain or leptomeningeal metastases
2. Patient is pre- or perimenopausal. Patient is pregnant or breast feeding or planning to become pregnant within five times the half-life of the IMPs after the end of treatment.
3. Patient has significant cardiovascular disease, such as cardiac disease (New York Heart Association Class II or greater), myocardial infarction or cerebrovascular accident within 6 months prior to initiation of study treatment, unstable arrhythmias, or unstable angina
4. Patient has other concomitant or previous malignancy, except adequately treated in-situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, cancer in complete remission for > 5 years
5. Patient has contraindication or shows hypersensitivity to the existing treatment with CDK4/6 inhibitor plus endocrine therapy
6. Patient shows evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the study medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results
7. Patient participated in another clinical study with an investigational medicinal product during the last 28 days before treatment initiation or 7 half-lives of previously used trial medication, whichever is longer or participate in such a study at the same time as this trial.

   Note: Participation in non-interventional clinical studies or registries is allowed.
8. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
9. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.
10. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate 12 months after randomization (PFS@12_stopping) | 12 months
  Proportion of patients alive and without progression according to radiologic imaging assessment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 54 months
  Time from randomization until progress
Time to treatment failure (TTF) | 54 months
  Time from randomization to end of treatment because of patient's wish, investigator's decision, toxicity, or progression
Progression-free survival (PFS2) | 54 months
  Time from re-treatment with CDK4/6 inhibitors to clinical disease progression or death from any cause
Time to treatment failure (TTF2) | 54 months
  Time to end of treatment because of patient's wish, investigator's decision, toxicity, or clinical progression after re-treatment with CDK4/6 inhibitors
Time to first use of chemotherapy | 54 months
  Time to first use of chemotherapy after progression on combined endocrine/CDK4/6 inhibitor treatment
Quality of life (QoL) EORTC QLQ-C30 | 54 months
  QoLassessed with the QoL questionnaire EORTC QLQ-C30
Quality of life (QoL) EORTC QLQ-BR23 | 54 months
  QoLassessed with the QoL questionnaire EORTC QLQ-BR23
Safety (rate of adverse events) | 54 months
  Type, incidence and severity of adverse events (AEs) and serious adverse events (SAEs) graded according to NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof., Study Director — Frankfurter Institut für Klinische Krebsforschung IKF GmbH
Locations (13):
- Germany (13):
  - Charité Berlin, Berlin
  - Hämatologische Onkologische Praxis im Medicum, Bremen
  - St. Johannes Hospital Dortmund, Dortmund
  - Praxis und Tagesklinik, Friedrichshafen
  - Hausärztliche und Onkologische Gemeinschaftspraxis, Gerlingen
  - Onkologische GP Gütersloh, Gütersloh
  - Hämatologisch-Onkologische Praxis Altona, Hamburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - MVZ für Hämatologie und Onkologie der MVZ Mülheim GmbH, Mülheim
  - MVZ für Hämatologie und Onkologie, Ravensburg
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Onkologisch-Gastroenterologische Schwerpunktpraxis Innere Medizin GbR, Singen
  - Onkologiezentrum Soest-Iserlohn, Soest

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared